CLINICAL TRIAL: NCT05227651
Title: Phase II Study on AK104 in Neoadjuvant Treatment of Cervical Cancer
Brief Title: AK104 in Neoadjuvant Treatment of Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-214
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 (Experimental): Patients will be treated with 1-4 cycles of neoadjuvant AK104. 2-4 weeks after the last cycle of neoadjuvant treatment, patients will undergo radical surgery.
  Interventions: Drug: AK104

INTERVENTIONS:
Drug: AK104 — IV infusion,Specified dose on specified days

SUMMARY:
Phase II open label study to evaluate the safety and efficacy of AK104 (anti-PD-1 and CTLA-4 bispecific antibody) in neoadjuvant treatment of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 & ≤75.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Histologically or cytologically confirmed diagnosis of primary cervical squamous cell carcinoma.
4. According to the 2018 International Federation of Cervical Cancer Obstetrics and Gynecology (FIGO) staging standard, the patient was diagnosed in stage IB2-IIA2.
5. Has not received any treatment before.
6. Has at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator.
7. Has adequate organ function.

Exclusion Criteria:

1. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
2. Active Hepatitis B or Hepatitis C.
3. History of severe bleeding tendency or coagulation disorder.
4. Undergone major surgery within 30 days prior to the first dose of study treatment.
5. Pregnant or lactating female patients.
6. Drug or alcohol abuse.
7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 6 mouths
  The number of participants experiencing an AE will be assessed. An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy.
Major pathological response (MPR) rate | within 14 working days after operation
  MPR rate is defined as the percentage of participants having ≤ 10% viable tumor cells in the pathological examination of resected specimens.

SECONDARY OUTCOMES:
R0 resection rate | within 14 working days after operation
  R0 resection rate is defined as the percentage of patients whose post-operative pathology indicate complete tumor resection with all margins being negative.
Pathological Complete Response (pCR) rate | within 14 working days after operation
  pCR rate is defined as the percentage of participants lacking of evidence of viable tumor cells in the pathological examination of resected specimens.
Objective response rates (ORR) | 4-6 weeks after the first cycle of neoadjuvant treatment
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hanzhong, Zhejiang, China